CLINICAL TRIAL: NCT01522430
Title: DENERVATION OF RENAL SYMPATHETIC ACTIVITY AND HYPERTENSION STUDY
Brief Title: Study of Catheter Based Renal Denervation Therapy in Hypertension
Acronym: DEPART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Jean Francois Argacha, Principal Investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140576
Record Dates: First submitted 2012-01-25; First posted 2012-01-31 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Resistant Hypertension; Renal Denervation; Ambulatory Blood Pressure; Renal Function
Keywords: Resistant hypertension; Renal denervation; Ambulatory blood pressure; Renal function; Simplicity catheter; Sham procedure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal angiography followed by renal sympathetic denervation (Experimental): Catheter based therapy for renal denervation using the Simplicity (TM) catheter (Ardian/Medtronic)
  Interventions: Procedure: Renal angiography followed by renal sympathetic denervation
- Renal angiography alone (Sham Comparator): Renal selective angiography using standardized method: Local anesthesia of the femoral site to allow the placement of a 4-Fr sheath in the femoral artery. Using JR-4 or similar diagnostic catheter, a selective renal angiography will be realized.
  Interventions: Procedure: Renal angiography alone

INTERVENTIONS:
Procedure: Renal angiography followed by renal sympathetic denervation — Radiofrequency catheter based therapy for renal denervation: Symplicity catheter will be advanced into the renal artery and connected to a radiofrequency generator. As previously described, four-to-six discrete, low-power radio frequency treatments will be applied along the length of both main renal arteries. At least four radiofrequency applications will be delivered in each renal artery, unless this is not feasible for anatomical reasons.
  Arms: Renal angiography followed by renal sympathetic denervation
Procedure: Renal angiography alone — Procedure will start with a local anesthesia of the femoral site to allow the placement of a 4-Fr sheath in the femoral artery, which allows a minimal risk of bleeding to the patient. Using JR-4 or similar diagnostic catheter, a selective renal angiography will be realized.
  Arms: Renal angiography alone

SUMMARY:
The DEPART study end points are to provide conclusive evidence, using a randomized, double blinded, sham procedure controlled study design, that radiofrequency renal denervation:

1. reduces daytime ambulatory blood pressure,
2. improves nocturnal dipping in blood pressure at the ambulatory blood pressure recording.

ELIGIBILITY:
Inclusion Criteria:

* They have a mandatory > 3 antihypertensive medication therapy, including a thiazide or a loop diuretic (according to the patient's renal function, unless documented side-effects) and at least one attempt to treat with spironolactone, given at usual recommended dose since at least 8 weeks, before inclusion,
* A mandatory check list of secondary cause of hypertension has been excluded
* They succeed the pill count test.
* They have a mandatory ambulatory blood pressure monitoring before inclusion with at least 70% of valid readings during daytime (08:00 am 08:00 pm, using a sampling frequency of 20 minutes, only devices validated according to http://www.dableducational.org are permitted), where daytime ambulatory blood pressure of systolic and/or diastolic blood pressure exceeds 135 mmHg and/or 85 mmHg, respectively. Daytime ambulatory blood pressure of systolic and/or diastolic blood pressure below 135 mmHg and/or 85 mmHg, respectively, is acceptable for inclusion in the study if the patient takes four or more antihypertensive medication (3).

Exclusion Criteria:

* Patients with an eGFR <30ml/min/m² are excluded,
* patients with known renal atherosclerotic lesions,
* previous procedures in the renal arteries,
* known unsuitable anatomy for the procedure,
* previous nephrectomy,
* contrast agent allergy,
* hyperthyroidia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
glomerular filtration rate | 6 month
  Isotopic and 24h urine sample measure of glomerular filtration rate.
Ambulatory systolic and diastolic blood pressure | 6 month
  Ambulatory systolic and diastolic blood pressure measured on 24h ABPM device

SECONDARY OUTCOMES:
Baroreflex sensitivity | 6 month
  Migroneugraphy recording of sympathetic nerve activity and testing of baroreflex sensitivity
Biological markers of acute kidney injury | baseline, H2, H6, 1, 3 and 6 months
  Urine sample for NGAL, L-FABP and Cystatine C at baseline, H2, H6, 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François ARGACHA, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium